CLINICAL TRIAL: NCT02993302
Title: Effects Of Oral Alfacalcidol On Maturation Of Dendritic Cells In Graves' Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Dyah Purnamasari, M.D., Ph.D, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSCM/FKUI
Record Dates: First submitted 2016-12-07; First posted 2016-12-15 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Graves Disease
Keywords: vitamin D; graves' disease; dendritic cells
MeSH Terms: conditions — Graves Disease | interventions — Calcitriol; alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTU-Oral 1α-D3 (Active Comparator): patients were given oral 1α-D3 at dose of 1.5 mcg once daily for 8 weeks in addition to propylthiouracil (PTU) 300 mg daily for 8 weeks as the treatment for Graves' disease with thyrotoxicosis
  Interventions: Drug: 1α-D3
- PTU-Placebos (Placebo Comparator): patients were given placebo tablets for 8 weeks in addition topropylthiouracil (PTU) 300 mg daily for 8 weeks as the treatment for Graves' disease with thyrotoxicosis
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 1α-D3 — patients were given PTU and 1α-D3
  Other Names: 1α 25-dihydroxyvitamin d3; alfacalcidol
  Arms: PTU-Oral 1α-D3
Drug: Placebos — patients were given PTU and placebos
  Other Names: placebo
  Arms: PTU-Placebos

SUMMARY:
Maturity level of dendritic cells (DC) plays a pivotal role in initiating and regulating autoimmunity. In Graves' disease (GD), DCs have more active immune responses than those in healthy subjects. Our previous study demonstrated immunoregulatory effects of in vitro 1,25-D3 on maturation of DC in GD patients. This study aims to evaluate the effect of oral 1α-D3 on DC maturation in GD patients.

DETAILED DESCRIPTION:
Patients with Graves' disease were divided into two groups: groups receiving oral 1α-D3 in addition to propylthiouracil (PTU) and groups receiving placebos in addition to PTU. Comparison of DC maturation were performed before and after the oral 1α-D3. DC maturation was assessed based on the expression of DC markers (HLA-DR, CD80, CD40, CD83, CD14 and CD206) and the ratio of cytokines interleukin-12/IL-10.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Graves' disease and still have not gone into remission
* Willing to participate in the research

Exclusion Criteria:

* Pregnant patient
* Suffered from severe liver disease
* Suffered from severe kidney disease
* Taking vitamin D substitution therapy
* Suffered from another autoimmune disease
* Suffered from malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dyah Purnamasari, M.D., Ph.D, Principal Investigator — Fakultas Kedokteran Universitas Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tamura M, Matsuura B, Miyauchi S, Onji M. Dendritic cells produce interleukin-12 in hyperthyroid mice. Eur J Endocrinol. 1999 Dec;141(6):625-9. doi: 10.1530/eje.0.1410625. PMID 10601966
- [Background] Banchereau J, Steinman RM. Dendritic cells and the control of immunity. Nature. 1998 Mar 19;392(6673):245-52. doi: 10.1038/32588. PMID 9521319
- [Background] Liang S, Ristich V, Arase H, Dausset J, Carosella ED, Horuzsko A. Modulation of dendritic cell differentiation by HLA-G and ILT4 requires the IL-6--STAT3 signaling pathway. Proc Natl Acad Sci U S A. 2008 Jun 17;105(24):8357-62. doi: 10.1073/pnas.0803341105. Epub 2008 Jun 11. PMID 18550825
- [Background] Inoue N, Watanabe M, Morita M, Tatusmi K, Hidaka Y, Akamizu T, Iwatani Y. Association of functional polymorphisms in promoter regions of IL5, IL6 and IL13 genes with development and prognosis of autoimmune thyroid diseases. Clin Exp Immunol. 2011 Mar;163(3):318-23. doi: 10.1111/j.1365-2249.2010.04306.x. Epub 2011 Jan 14. PMID 21235536
- [Background] Khalilzadeh O, Anvari M, Esteghamati A, Momen-Heravi F, Mahmoudi M, Rashidi A, Amiri HM, Ranjbar M, Tabataba-Vakili S, Amirzargar A. The interleukin-1 family gene polymorphisms and Graves' disease. Ann Endocrinol (Paris). 2010 Sep;71(4):281-5. doi: 10.1016/j.ando.2010.01.005. Epub 2010 Apr 18. PMID 20400062
- [Background] Croizet K, Rabilloud R, Kostrouch Z, Nicolas JF, Rousset B. Culture of dendritic cells from a nonlymphoid organ, the thyroid gland: evidence for TNFalpha-dependent phenotypic changes of thyroid-derived dendritic cells. Lab Invest. 2000 Aug;80(8):1215-25. doi: 10.1038/labinvest.3780129. PMID 10950112
- [Background] Dedecjus M, Stasiolek M, Brzezinski J, Selmaj K, Lewinski A. Thyroid hormones influence human dendritic cells' phenotype, function, and subsets distribution. Thyroid. 2011 May;21(5):533-40. doi: 10.1089/thy.2010.0183. Epub 2010 Dec 29. PMID 21190445
- [Background] Hughes GC, Clark EA. Regulation of dendritic cells by female sex steroids: relevance to immunity and autoimmunity. Autoimmunity. 2007 Sep;40(6):470-81. doi: 10.1080/08916930701464764. PMID 17729041
- [Background] Duperrier K, Farre A, Bienvenu J, Bleyzac N, Bernaud J, Gebuhrer L, Rigal D, Eljaafari A. Cyclosporin A inhibits dendritic cell maturation promoted by TNF-alpha or LPS but not by double-stranded RNA or CD40L. J Leukoc Biol. 2002 Nov;72(5):953-61. PMID 12429717
- [Background] Berer A, Stockl J, Majdic O, Wagner T, Kollars M, Lechner K, Geissler K, Oehler L. 1,25-Dihydroxyvitamin D(3) inhibits dendritic cell differentiation and maturation in vitro. Exp Hematol. 2000 May;28(5):575-83. doi: 10.1016/s0301-472x(00)00143-0. PMID 10812248
- [Background] Wahono CS, Rusmini H, Soelistyoningsih D, Hakim R, Handono K, Endharti AT, Kalim H, Widjajanto E. Effects of 1,25(OH)2D3 in immune response regulation of systemic lupus erithematosus (SLE) patient with hypovitamin D. Int J Clin Exp Med. 2014 Jan 15;7(1):22-31. eCollection 2014. PMID 24482685
- [Background] Bartels LE, Jorgensen SP, Bendix M, Hvas CL, Agnholt J, Agger R, Dahlerup JF. 25-Hydroxy vitamin D3 modulates dendritic cell phenotype and function in Crohn's disease. Inflammopharmacology. 2013 Apr;21(2):177-86. doi: 10.1007/s10787-012-0168-y. Epub 2013 Jan 23. PMID 23341164
- [Background] Agmon-Levin N, Theodor E, Segal RM, Shoenfeld Y. Vitamin D in systemic and organ-specific autoimmune diseases. Clin Rev Allergy Immunol. 2013 Oct;45(2):256-66. doi: 10.1007/s12016-012-8342-y. PMID 23238772
- [Background] Zhou H, Xu C, Gu M. Vitamin D receptor (VDR) gene polymorphisms and Graves' disease: a meta-analysis. Clin Endocrinol (Oxf). 2009 Jun;70(6):938-45. doi: 10.1111/j.1365-2265.2008.03413.x. Epub 2008 Sep 8. PMID 18782354
- [Background] Budiyati AD, Setiyono A, Tarigan E and Wibowo H. The effect of alpha fetoprotein on NF-kB translocation in lipopolysaccharide induced monocyte-derived dendritic cell. Med J Indones. 2012; 21.
- [Background] Hewison M. Vitamin D and the immune system: new perspectives on an old theme. Endocrinol Metab Clin North Am. 2010 Jun;39(2):365-79, table of contents. doi: 10.1016/j.ecl.2010.02.010. PMID 20511058
- [Background] Antico A, Tampoia M, Tozzoli R, Bizzaro N. Can supplementation with vitamin D reduce the risk or modify the course of autoimmune diseases? A systematic review of the literature. Autoimmun Rev. 2012 Dec;12(2):127-36. doi: 10.1016/j.autrev.2012.07.007. Epub 2012 Jul 7. PMID 22776787
- [Background] Hunt PJ, Marshall SE, Weetman AP, Bell JI, Wass JA, Welsh KI. Cytokine gene polymorphisms in autoimmune thyroid disease. J Clin Endocrinol Metab. 2000 May;85(5):1984-8. doi: 10.1210/jcem.85.5.6588. PMID 10843185
- [Result] Bartels LE, Bendix M, Hvas CL, Jorgensen SP, Agnholt J, Agger R, Dahlerup JF. Oral vitamin D3 supplementation reduces monocyte-derived dendritic cell maturation and cytokine production in Crohn's disease patients. Inflammopharmacology. 2014 Apr;22(2):95-103. doi: 10.1007/s10787-013-0197-1. Epub 2013 Dec 29. PMID 24374976
- [Result] Bartosik-Psujek H, Tabarkiewicz J, Pocinska K, Stelmasiak Z, Rolinski J. Immunomodulatory effects of vitamin D on monocyte-derived dendritic cells in multiple sclerosis. Mult Scler. 2010 Dec;16(12):1513-6. doi: 10.1177/1352458510379611. Epub 2010 Aug 25. PMID 20739336
- [Result] Abou-Raya A, Abou-Raya S, Helmii M. The effect of vitamin D supplementation on inflammatory and hemostatic markers and disease activity in patients with systemic lupus erythematosus: a randomized placebo-controlled trial. J Rheumatol. 2013 Mar;40(3):265-72. doi: 10.3899/jrheum.111594. Epub 2012 Dec 1. PMID 23204220 (Retraction: PMID 30504482 J Rheumatol. 2018 Dec;45(12):1713)
- [Result] Pani MA, Regulla K, Segni M, Hofmann S, Hufner M, Pasquino AM, Usadel KH, Badenhoop K. A polymorphism within the vitamin D-binding protein gene is associated with Graves' disease but not with Hashimoto's thyroiditis. J Clin Endocrinol Metab. 2002 Jun;87(6):2564-7. doi: 10.1210/jcem.87.6.8562. PMID 12050214
- [Result] Yasuda T, Okamoto Y, Hamada N, Miyashita K, Takahara M, Sakamoto F, Miyatsuka T, Kitamura T, Katakami N, Kawamori D, Otsuki M, Matsuoka TA, Kaneto H, Shimomura I. Serum vitamin D levels are decreased in patients without remission of Graves' disease. Endocrine. 2013 Feb;43(1):230-2. doi: 10.1007/s12020-012-9789-6. Epub 2012 Sep 15. No abstract available. PMID 22983830
- [Result] Kawakami-Tani T, Fukawa E, Tanaka H, Abe Y, Makino I. Effect of 1 alpha-hydroxyvitamin D3 on serum levels of thyroid hormones in hyperthyroid patients with untreated Graves' disease. Metabolism. 1997 Oct;46(10):1184-8. doi: 10.1016/s0026-0495(97)90214-6. PMID 9322804
- [Result] D Purnamasari PS, S Djauzi, S Setiati, A Harahap, J Prihartono. Effects of In Vitro 1,25 Dihydroxyvitamin D on Maturation of Dendritic Cells in Graves' Disease Patients. Asian J Pharm Clin Res. 2016; 9: 221-4
- [Result] Handono K, Gani AA, Ekawati M and Wahono S. Serum level of vitamin D and autoantibodies level in systemic lupus erythematosus (SLE) patients. Journal of Pharmacy and Biological Sciences. 2012; 3: 16-20
- [Result] Tamaru M, Matsuura B, Onji M. Increased levels of serum interleukin-12 in Graves' disease. Eur J Endocrinol. 1999 Aug;141(2):111-6. doi: 10.1530/eje.0.1410111. PMID 10427152
- [Result] D Purnamasari PS, S Djauzi. Sunlight-derived vitamin D affects interleukin-4 level, T helper 2 serum cytokines, in patients with Graves' disease: a prospective cohort study. Med J Indones. 2015; 24: 228-33

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2014 - May 2015, Patients with Graves' disease who are still in hyperthyroid condition at the outpatient clinic of Endocrinology Department of Dr. Cipto Mangunkusumo Hospital in Jakarta, Indonesia.
Groups:
- PTU + Oral 1α-D3: patients were given oral 1α-D3 at dose of 1.5 mcg once daily for 8 weeks in addition to propylthiouracil (PTU) 300 mg daily for 8 weeks as the treatment for Graves' disease with thyrotoxicosis
  1α-D3: patients were given PTU and 1α-D3
- PTU + Placebos: patients were given placebo tablets for 8 weeks in addition topropylthiouracil (PTU) 300 mg daily for 8 weeks as the treatment for Graves' disease with thyrotoxicosis
  Placebos: patients were given PTU and placebos
Period: Overall Study
Arm/Group | PTU + Oral 1α-D3 | PTU + Placebos
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTU + Oral 1α-D3 | PTU + Placebos | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.67 (7.92) | 38.15 (9.34) | 36 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 2 | 0 | 2
Duration of illness [Median (Full Range); unit: months] | 18 [2 to 266] | 27 [2 to 204] | 24 [2 to 266]
thyroid-stimulating hormone (TSH) levels [Median (Inter-Quartile Range); unit: µIU/l] | 0.01 [0.01 to 1.86] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 1.86]
free thyroxine (fT4) levels [Median (Full Range); unit: ng/dL] | 6.9 [2.95 to 7.77] | 4.2 [2.51 to 7.77] | 5.04 [2.51 to 7.77]
TSH receptor antibody (TRAb) levels [Median (Full Range); unit: U/L] | 14.46 [3.42 to 87.74] | 9.55 [3.3 to 55.4] | 14.174 [3.3 to 87.74]
Ca ion levels [Mean (Standard Deviation); unit: mmol/L] | 1.13 (0.05) | 1.13 (0.06) | 1.13 (0.05)
Vitamin 25-D3 levels [Mean (Standard Deviation); unit: ng/mL] | 24.4 (7.81) | 25.55 (5.56) | 25 (6.62)

OUTCOME MEASURES:

1. Primary Outcome: CD80 Level
Description: Dendritic cells maturation levels were measured by the CD80 (cluster of differentiation 80)
Time Frame: 1 year
Measure: Median (Full Range); unit: nM
Arm/Group | PTU + Oral 1α-D3 | PTU + Placebos
Number analyzed (Participants) | 13 | 12
nM | 45.60 [31.20 to 139.36] | 54.51 [39.47 to 69.55]
Statistical Analysis 1: Comparison: PTU + Oral 1α-D3 vs PTU + Placebos; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney)

2. Primary Outcome: CD206 Level
Description: Dendritic cells maturation levels were measured by the CD206
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | PTU + Oral 1α-D3 | PTU + Placebos
Number analyzed (Participants) | 13 | 12
nM | 54.08 (23.46) | 53.42 (13.72)
Statistical Analysis 1: Comparison: PTU + Oral 1α-D3 vs PTU + Placebos; Test type: Other; p = 0.47, Wilcoxon (Mann-Whitney)

3. Primary Outcome: IL-12/IL-10 Ratio
Description: Dendritic cells maturation levels were measured by the IL-12 (interleukin-12)/IL-10 ratio
Time Frame: 1 year
Measure: Median (Full Range); unit: ratio
Arm/Group | PTU + Oral 1α-D3 | PTU + Placebos
Number analyzed (Participants) | 13 | 12
ratio | 0.49 [0.04 to 8.01] | 0.21 [0.03 to 3.40]
Statistical Analysis 1: Comparison: PTU + Oral 1α-D3 vs PTU + Placebos; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney)

4. Primary Outcome: fT4 Levels
Description: fT4 (free thyroxine)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | PTU + Oral 1α-D3 | PTU + Placebos
Number analyzed (Participants) | 13 | 12
ng/dL | 2.65 (2.06) | 2.09 (1.19)

ADVERSE EVENTS:
Arm/Group | PTU + Oral 1α-D3 | PTU + Placebos
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes